CLINICAL TRIAL: NCT00578890
Title: Comparison of Medical and Medical-surgical Management of Diabetic Foot Osteomyelitis
Brief Title: a Randomized Controlled Trial Comparing Medical and Medical-surgical Treatment in Diabetic Foot Osteomyelitis
Acronym: DIPIOS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: not enough recruitment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Mathieu QUINTIN, Delegation of clinical research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060218
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2011-06

CONDITIONS: Diabetic Foot
Keywords: diabetic foot; osteomyelitis
MeSH Terms: conditions — Diabetic Foot; Osteomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Medical/surgical treatment versus medical treatment

INTERVENTIONS:
Procedure: Medical/surgical treatment versus medical treatment — A 12 week course antibiotics versus a limited resection of infected bone associated with a 4 week course antibiotics.

SUMMARY:
Osteomyelitis is a frequent complication of diabetic foot ulcer. Several therapeutic strategies are used : medical treatment with antibiotics and foot offloading or surgical treatment consisting in the resection of infected bone and a shorter antibiotic course. The medical treatment risk is a longer healing time and a risk of bone infection relapse. The surgical treatment risk is the ulcer relapse because of the modification of the foot structure. These treatments need to be compared in terms of benefit/risk ratio. Our hypothesis is : 1) in the medical treatment group a 7 month mean healing time of and a 15% osteomyelitis recurrence rate;2) in the medical-surgical treatment group a 4 month mean healing time and a 10% osteomyelitis recurrence rate.

DETAILED DESCRIPTION:
The study aim is to compare the rate of therapeutic success of the secondary ostéite with a wound of the foot diabetic, obtained either by a single medical coverage(care), or by a medical surgical coverage(care). The therapeutic success being defined by the association of 1) the absence of local distribution(broadcasting) of the ostéite 2) the healing of the wound 3) in 12 months of the healing the absence of local recurrence of the ostéite

ELIGIBILITY:
Inclusion Criteria:

* diabetes
* neuropathy and a forefoot ulcer
* osteomyelitis on X ray involving one or two contiguous ray
* confirmed osteomyelitis on bone biopsy if a metatarsal head is involved
* palpable distal pulses

Exclusion Criteria:

* glomerular filtration rate < 30ml/min
* whole bone destruction
* contra-indication for off loading
* ASAT or ALAT > three times normal rate
* immunosuppressive drugs
* Charcot foot on the concerned foot
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
no osteomyelitis spreading and wound healing and no osteomyelitis relapse 12 months after wound healing | 12 months after healing

SECONDARY OUTCOMES:
amputation rate | before healing
healing time | end of study
ulcer relapse 12 months after healing | 12 months after healing

CONTACTS AND LOCATIONS:
Overall Officials: Agnès Hartemann-Heurtier, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris